CLINICAL TRIAL: NCT05366517
Title: Evaluation of Repeating Low-intensity Shockwave Therapy (LiST) for Refractory Non-bacterial Prostatitis/Pelvic Pain Syndrome: a Single Arm Prospective Study
Brief Title: Repeating LiST for Refractory Non-bacterial Prostatitis/Pelvic Pain Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute for the Study of Urological Diseases, Greece (Other)
Responsible Party: Principal Investigator, Dimitrios Hatzichristou, Professor, Institute for the Study of Urological Diseases, Greece
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMOP CPPS
Record Dates: First submitted 2022-05-04; First posted 2022-05-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Chronic Prostatitis With Chronic Pelvic Pain Syndrome
MeSH Terms: conditions — Prostatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group (Other): LiST active treatment group
  Interventions: Device: Dornier Aries 2 device

INTERVENTIONS:
Device: Dornier Aries 2 device — For 6 weeks, patients will receive 6 sessions with active LiST probe, 2 session per week. The ARIES 2 device by Dornier will be used with a treatment protocol: 5000 SW, energy flux density = 0.096 mJ/mm2 (energy level 7) frequency = 5Hz

SUMMARY:
The aim of the study is to investigate the efficacy and safety of LiST retreatment for CP/CPPS patients.A total of 50 patients with CP/CPPS diagnosis who were previously treated with 6 sessions of LiST will participate in this study.The primary study parameter is the CP/CPPS-related pain complaints and it will be assessed by the NIH-CPSI

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be between 18-60 years of age.
2. Participant has signed and dated the appropriate Informed Consent document.
3. Participant has had a clinical diagnosis of CP/CPPS defined as symptoms of discomfort or pain in the perineal or pelvic region for at least a three (3) month period within the last six (6) months.
4. Participant has received 6 sessions (1/week or 2/week, energy level 7, Dornier ARIES 2) of LIST the last 12 months for the treatment of CP/CPPS reporting amelioration but without complete remission of CP/CPPS symptoms ( at over 1 UPOINT positive domain).

Exclusion Criteria:

1. Participant has evidence of facultative Gram negative or enterococcus with a value of ≥ 1000 CFU/ml in mid-stream urine (VB2).
2. Participant has a history of prostate, bladder or urethral cancer.
3. Participant has undergone pelvic radiation or systemic chemotherapy.
4. Participant has undergone intravesical chemotherapy.
5. Participant has unilateral orchialgia without pelvic symptoms, active urethral stricture or bladder stones, or any other urological condition associated with LUTS, any neurological disease or disorder affecting the bladder.
6. Participant has undergone prostate surgery or treatment.
7. Participant with penile or urinary sphincter implants.
8. Participant has been diagnosed with cancer during the last 5 years, or had any surgery in the pelvis.
9. Participant has a neurological impairment or psychiatric disorder preventing his understanding of consent and his ability to comply with the protocol.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The change of the pain domain of NIH-CPSI score from baseline to 12 weeks after final treatment. | from baseline to 12 weeks after final treatment.
  CP/CPPS-related complaints will be assessed by the the National Institutes of Health Chronic Prostatitis Symptom Index (NIH-CPSI). The questionnaire designed to provide symptom scores for patients with chronic prostatitis. The index provides scores on pain (items 1-4), urinary symptoms (items 5-6), and quality of life (items 7-9).Total score ranges from 0 to 35 (higher values represent worse outcome).The index provides a special pain domain (items 1-4) and the score for this domain ranges from 0 to 21.

SECONDARY OUTCOMES:
The change of the pain domain of NIH-CPSI score from baseline to 4 weeks after final treatment. | from baseline to 4 weeks after final treatment.
  CP/CPPS-related complaints will be assessed by the the National Institutes of Health Chronic Prostatitis Symptom Index (NIH-CPSI). The questionnaire designed to provide symptom scores for patients with chronic prostatitis. The index provides scores on pain (items 1-4), urinary symptoms (items 5-6), and quality of life (items 7-9).Total score ranges from 0 to 35 (higher values represent worse outcome).The index provides a special pain domain (items 1-4) and the score for this domain ranges from 0 to 21.
The change of total NIH-CPSI score (Q1-9)from baseline to 4 and 12 weeks after final treatment | baseline, 4 and 12 weeks after final treatment
  CP/CPPS-related complaints will be assessed by the the National Institutes of Health Chronic Prostatitis Symptom Index (NIH-CPSI). The questionnaire designed to provide symptom scores for patients with chronic prostatitis. The index provides scores on pain (items 1-4), urinary symptoms (items 5-6), and quality of life (items 7-9).Total score ranges from 0 to 35 (higher values represent worse outcome).
The change of urinary symptoms (Q 5-6) and quality of life domains (Q 7-9) of the NIH-CPSI score from baseline to 4 and 12 weeks after final treatment | baseline, 4 and 12 weeks after final treatment
  CP/CPPS-related complaints will be assessed by the the National Institutes of Health Chronic Prostatitis Symptom Index (NIH-CPSI). The questionnaire designed to provide symptom scores for patients with chronic prostatitis. The index provides scores on pain (items 1-4), urinary symptoms (items 5-6), and quality of life (items 7-9).Total score ranges from 0 to 35 (higher values represent worse outcome).The index provides a special urinary symptom domain (items 5-6) and the score for this domain ranges from 0 to 10.
The change of quality of life domains (Q 7-9) of the NIH-CPSI score from baseline to 4 and 12 weeks after final treatment | baseline, 4 and 12 weeks after final treatment
  CP/CPPS-related complaints will be assessed by the the National Institutes of Health Chronic Prostatitis Symptom Index (NIH-CPSI). The questionnaire designed to provide symptom scores for patients with chronic prostatitis. The index provides scores on pain (items 1-4), urinary symptoms (items 5-6), and quality of life (items 7-9).Total score ranges from 0 to 35 (higher values represent worse outcome).The index provides a special urinary symptom domain (items 5-6) and the score for this domain ranges from 0 to 10.
The change of IIEF-ED score from baseline to 4 and 12 weeks after final treatment | baseline, 4 and 12 weeks after final treatment
  It will be assessed by International Index of Erectile Function -Erectile Domain (IEF-ED) score. A questionnaire designed to evaluate erectile capabilities. The questionnaire provides a score between 5 and 30.The severity categories are: 1-10 severe ED, 10-16 moderate ED, 17-21 moderate to mild ED, 22-25 mild ED, 26-30 no ED
The difference between the LiST and sham group in the change of UPPOINTS phenotype- number of positive domainsfrom baseline to 4 and 12 weeks after final | baseline, 4 and 12 weeks after final treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Hatzichristou, Professor, Principal Investigator — Institute for the Study of Urological Diseases, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No